CLINICAL TRIAL: NCT02661334
Title: Measuring Uniformed Servicemembers' Fitness Scores on Creatine Loading and Exercise (MUSSCLE)
Brief Title: Measuring Uniformed Servicemembers' Fitness Scores on Creatine Loading and Exercise
Acronym: MUSSCLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FDG20150021H
Record Dates: First submitted 2015-12-07; First posted 2016-01-22 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Physical Fitness
Keywords: creatine; creatine monohydrate; supplement; exercise; fitness
MeSH Terms: conditions — Motor Activity | interventions — Creatine; Flour

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 30g white rice flour
  Interventions: Dietary Supplement: Rice Flour
- Low dose (Experimental): 5g/day Creatine Monohydrate (25g white rice flour) for 28 days
  Interventions: Dietary Supplement: Creatine Monohydrate; Dietary Supplement: Rice Flour
- Loading dose (Experimental): Creatine Monohydrate 20g/day (10g white rice flour) for 7 days, followed by maintenance dose of Creatine Monohydrate 5g/day (25g white rice flour) for the remaining 21 days
  Interventions: Dietary Supplement: Creatine Monohydrate; Dietary Supplement: Rice Flour
- High dose (Experimental): High dose of Creatine Monohydrate 20g/day (10g white rice flour) for the entire 28 day period
  Interventions: Dietary Supplement: Creatine Monohydrate; Dietary Supplement: Rice Flour

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate — Creatine monohydrate is a very common supplement used by enthusiasts, athletes, and the general populace
  Arms: High dose; Loading dose; Low dose
Dietary Supplement: Rice Flour — rice flour powder matched for color, appearance, taste, and solubility

SUMMARY:
The purpose of this study is to compare the physical fitness performance-as measured by the Air Force Physical Fitness Test (PFT)-of subjects that, in conjunction with exercise, will take creatine supplementation over a four week period versus those that do not.

DETAILED DESCRIPTION:
The purpose of this study is to compare the physical fitness performance-as measured by the Air Force Physical Fitness Test (PFT)-of subjects that, in conjunction with exercise, will take creatine supplementation over a four week period versus those that do not. Based on the literature, there is evidence to support that creatine supplementation may increase available levels of muscle phosphocreatine (PCr), an important energy reservoir that is initially expended with intense muscular contraction and then regenerated during episodes of rest. While mechanistically plausible, the effects of creatine on the specific measures of the PFT (push-ups, sit-ups, 1.5 mile run, and abdominal circumference) have not been evaluated. The target population is Active Duty Air Force (ADAF) service members who perform perform the PFT. As such, this represents a population with occupational requirements to maintain their fitness at a designated level. If short-term creatine supplementation does help to improve PFT scores, trainers, commanders, and unit physicians may wish to consider recommending its use. While generally considered safe, additional data will also be collected to evaluate both the qualitative and quantitative side-effects of creatine supplementation over the study period. If the hypothesis is correct and creatine supplementation is shown to be both effective and safe, additional studies may be warranted to evaluate its impact on ADAF service members who have failed the PFT and/or are at risk of being separated from the AF for unsatisfactory fitness performance. In short, this study has the potential to dramatically affect the recommendations and practices of ADAF service members related to use of creatine supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age ≥18
* Willing to exercise five days per week for four weeks, performing each component of the AF PFT at least once per week
* Willing to adhere to a prescribed supplementation regimen, including spaced dosing two times per day
* Able to meet all study follow-up and testing requirements as outlined in section 6.4 of this protocol

Exclusion Criteria:

* History of:
* Chronic kidney dysfunction
* Liver failure
* Rhabdomyolysis
* Compartment syndrome
* Current
* Pregnancy
* Musculoskeletal injury
* Fitness exemption from any component of the AF PFT (e.g. AF 469, "profile")
* Kidney injury
* Diabetes
* Hypertension, requiring medication
* Allergy to rice
* Admission to the hospital within the past 30 days
* Creatine supplementation within the past 90 days

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Determine the effect of creatine supplementation on anaerobic performance in the PFT by measuring change in repetitions of push-ups and sit-ups. | 28 days
  An initial mock AF PFT will be administered. Individual component raw numbers, scores, and composite scores will be recorded. Participants will self-take their prescribed regimen twice a day, in addition to exercise 5 days/week. Within 7 days of completing the prescribed treatment and exercise course, participants will undergo another mock AF PFT. The individual component raw numbers, scores, and composite scores will be recorded and compared to initial mock scores
Determine the effect of creatine supplementation on aerobic performance in the PFT by measuring change in 1.5 mile run time. | 28 days
  An initial mock AF PFT will be administered. Individual component raw numbers, scores, and composite scores will be recorded. Participants will self-take their prescribed regimen twice a day, in addition to exercise 5 days/week. Within 7 days of completing the prescribed treatment and exercise course, participants will undergo another mock AF PFT. The individual component raw numbers, scores, and composite scores will be recorded and compared to initial mock scores
Determine the effect of creatine supplementation on body composition as it relates to the PFT by measuring change in abdominal circumference | 28 days
  An initial mock AF PFT will be administered. Individual component raw numbers, scores, and composite scores will be recorded. Participants will self-take their prescribed regimen twice a day, in addition to exercise 5 days/week. Within 7 days of completing the prescribed treatment and exercise course, participants will undergo another mock AF PFT. The individual component raw numbers, scores, and composite scores will be recorded and compared to initial mock scores

SECONDARY OUTCOMES:
Determine how renal function is affected by creatine supplementation by measuring renal function labs (BUN/Creatinine/GFR-with Cys C) before and after the study period. | 28 days
  Labs will be draw before initiation of prescribed treatment. Once the 28-day study period has been completed, each participant will be sent to the DGMC laboratory for a final blood draw
Assess for possible liver damage resulting from creatine supplementation by measuring liver function labs (AST/ALT/Alk Phos) before and after the study period. | 28 days
  Labs will be draw before initiation of prescribed treatment. Once the 28-day study period has been completed, each participant will be sent to the DGMC laboratory for a final blood draw
Evaluate the risk of rhabdomyolysis with creatine supplementation by measuring creatine kinase before and after the study period. | 28 days
  Labs will be draw before initiation of prescribed treatment. Once the 28-day study period has been completed, each participant will be sent to the DGMC laboratory for a final blood draw
Treatment compliance as determined by medication diary. | 28 days
  Participants will be given a log book to record their supplement compliance. They will meet with the study coordinator at the two-week mark (between days 10-14) and review their logbook to ensure they are appropriately taking their supplements. Once the 28-day study period has been completed, each participant with meet with a study team member again to turn in their log book
Quality of workout as determined by exercise diary. | 28 days
  Participants will be given a log book to record their exercise history. They will meet with the study coordinator at the two-week mark (between days 10-14) and review their logbook to ensure they are meeting the requirement of exercising 4 out of 5 days/week. Once the 28-day study period has been completed, each participant with meet with a study team member again to turn in their log book

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Kasteler, MD, Principal Investigator — US Air Force
Locations (1):
- David Grant Medical Center, Fairfield, California, United States

IPD SHARING:
Plan to Share IPD: No